CLINICAL TRIAL: NCT05357456
Title: A Single Center, Prospective, Observational Study to Explore and Evaluate the Differences of Cognitive Function and Brain Function Between Non-functioning Adrenal Adenomas and Autonomous Cortisol Secretion Patients, and the Different Treatments Methods on Cognitive Function and Brain Function in Patients With Autonomous Cortisol Secretion
Brief Title: Performances on Cognitive Functions and Brain Function and Follow-up After Different Treatments in Patients With Autonomous Cortisol Secretion: a Single-center, Prospective, Observational Study
Status: Recruiting | Type: Observational
Sponsor: The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other)
Responsible Party: Principal Investigator, Dalong Zhu, Chief Physician, The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School
Other Study IDs: LP2022
Record Dates: First submitted 2022-04-27; First posted 2022-05-02 (Actual); Last update posted 2022-05-02 (Actual); Status verified 2022-04

CONDITIONS: Autonomous Cortisol Secretion; Adrenal Incidentaloma; Non-functioning Adrenal Adenomas
Keywords: cognitive function; functional MRI; treatment
MeSH Terms: conditions — Adrenal incidentaloma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- autonomous cortisol secretion: Patients admitted to the hospital with adrenal incidentalomas are evaluated for adrenal function, and then ACS patients are diagnosed based on the serum cortisol ≥ 50 nmol/L following the 1 mg dexamethasone suppression test and without any other signs or symptoms of cortisol excess.Patients with ACS will undergo a physical exam, cognitive function test as well as structural and functional brain MRI at baseline and 12 months after their surgery or conservative treatment.
  Interventions: Behavioral: Cognitive function assessment; functional magnetic resonance imaging; Procedure: laparoscopic adrenal surgery
- non-functioning adrenal adenomas: Patients admitted to the hospital with adrenal incidentalomas are evaluated for adrenal function, and then non-functioning adrenal adenomas patients are diagnosed based on the serum cortisol < 50 nmol/L following the 1 mg dexamethasone suppression test .Patients with non-functioning adrenal adenomas will undergo a physical exam, cognitive function test as well as structural and functional brain MRI at baseline.
  Interventions: Behavioral: Cognitive function assessment; functional magnetic resonance imaging

INTERVENTIONS:
Behavioral: Cognitive function assessment; functional magnetic resonance imaging — cognitive function measurement
  Other Names: fMRI
Procedure: laparoscopic adrenal surgery — Only a subgroup of the autonomous cortisol secretion patients will have the laparoscopic adrenal surgery
  Groups: autonomous cortisol secretion

SUMMARY:
This is a single center, prospective, observational study to explore and evaluate the differences on cognitive function and brain function by functional-MRI in autonomous cortisol secretion patients, and the different treatments methods on the cognitive function and brain function in patients with autonomous cortisol secretion

DETAILED DESCRIPTION:
Glucocorticoids, mainly cortisol, play a crucial role in the allostatic process of adjustment to stressors and can determine important changes in central nervous system structures. It is well known that Cushing's syndrome (CS) is associated with neurocognitive impairment in about two-thirds of cases. In CS the most frequent reported alterations are memory impairment (about 83% of cases) and reduced concentration (66% of cases) . Unfortunately, these alterations are only partially reversible after the hypercortisolism resolution. As so far, data related to the impact of autonomous cortisol secretion (ACS) on cognitive function are scarce and lack of magnetic resonance indicators. Few studies have studied the cognitive function changes of patients with ACS by surgical and conservative treatment. In the single center, prospective and observational study we aim to explore cognitive functions and brain function by functional-MRI in adrenal incidentaloma patients in relation to the presence of ACS and, secondly, in a group of acs patients, the effect of adrenalectomy on cognitive functions and brain function.

ELIGIBILITY:
Inclusion Criteria:

* age 20-65 years;
* ≥ 6 years of education；
* right-handed;
* complete entire cognitive function tests;
* adrenal lesions ≥ 1 cm in diameter;
* patients with non-functioning adrenal adenomas;
* patients with autonomous cortisol secretion.

Exclusion Criteria:

* < 6 years of education;
* age < 20 years or > 65 years;
* maximum diameter of AI <1cm;
* active malignancies;
* with a history of thyroid disease;
* with a history of acute infection in the last month;
* central nervous system diseases, including brain trauma, intracranial hemorrhage, acute cerebral infarction, etc;
* contraindications of MRI examination: such as implantation of metal prosthesis in vivo, claustrophobia, etc;
* adrenal tuberculosis;
* suspected or diagnosed adrenocortical carcinoma;
* unable to complete entire cognitive function tests;
* current use of steroids or any drugs known to alter steroid synthesis or metabolism in the previous 3 months;
* clinical Cushing syndrome;
* Cushing disease;
* primary hyperaldosteronism;
* pheochromocytoma;
* severe impairment of heart, liver, kidney and other organs;
* pregnant and lactating women

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: autonomous cortisol secretion and non-functioning adrenal adenomas patients
Sampling Method: Probability Sample
Enrollment: 62 (Estimated)
Dates: Start 2021-10-01 (Actual); Primary Completion 2024-10-01 (Estimated); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
Participants' personal information | 1 day
  Self-reported information(education in years)
Physical assessments | 1 day
  BMI(body mess index) in kg/m^2
Imaging examinations | 1 day
  Adrenal adenoma size in cm
Montreal Cognitive Assessment (MoCA) | 20 minutes
  The MoCA is a Global cognitive screening test designed to assist Health Professionals in detection of mild cognitive impairment.
Mini-Mental State Examination (MMSE) | 20 minutes
  The MMSE is a cognitive screening test designed to assist Health Professionals in detection of mild cognitive impairment.
Repeatable Battery for the Assessment of Neuropsychological Status (RBANS) | 1 hour
  The RBANS is a cognitive screening test designed to assist Health Professionals in evaluation of multiple cognitive subdomains
Rest Functional MRI of the brain function. | 40 minutes
  Rs-fMRI
Screening for adrenal cortisol hypersecretion | 1 day
  Patients were given 1 mg dexamethasone orally at 24:00 am, and the cortisol levels were measured at 8:00 am the following morning

SECONDARY OUTCOMES:
Changes from basline global cognitive functions | 12 months after the laparoscopic adrenal surgery (for patients with autonomous cortisol secretion who are willing to operate)]
  MoCA
Changes from basline multiple cognitive subdomains | 12 months after the laparoscopic adrenal surgery (for patients with autonomous cortisol secretion who are willing to operate)]
  RBANS
Change from baseline Functional magnetic resonance imagine | 12 months after the laparoscopic adrenal surgery (for patients with autonomous cortisol secretion who are willing to operate)]
  Rs-fMRI
Changes from basline global cognitive functions | 12 months after the conservative treatment (for patients with autonomous cortisol secretion who are not willing to operate)]
  MoCA
Changes from basline multiple cognitive subdomains | 12 months after the conservative treatment (for patients with autonomous cortisol secretion who are not willing to operate)]
  RBANS
Change from baseline Functional magnetic resonance imagine | 12 months after the conservative treatment (for patients with autonomous cortisol secretion who are not willing to operate)]
  Rs-fMRI

CONTACTS AND LOCATIONS:
Overall Officials: Dalong Zhu, MD,PhD, Principal Investigator — The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School
Locations (1):
- Department of Endocrinology, Drum Tower Hospital affiliated to Nanjing University Medical School, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Liu MS, Tian ZY, Zhang Z, Yang F, Lou Y, Wang YJ, Zeng YJ, Zhang ZW, Zhu DL, Li P. Impaired Cognitive Function in Patients With Autonomous Cortisol Secretion in Adrenal Incidentalomas. J Clin Endocrinol Metab. 2023 Feb 15;108(3):633-641. doi: 10.1210/clinem/dgac603. PMID 36263685